CLINICAL TRIAL: NCT00419796
Title: A 4-Week, Multicentre, Randomized, Double-Blind, Placebo Controlled, Double Dummy, Parallel Group Study, to Assess the Effect of Lumiracoxib 100 mg o.d. and Ibuprofen 600 mg t.i.d on 24-Hour Blood Pressure Profile and on Urinary Excretions of Eicosanoids, in Osteoarthritis Patients With Controlled Hypertension
Brief Title: Effects of Lumiracoxib and Ibuprofen on Blood Pressure and Urinary Eicosanoid Excretion in Osteoarthritis Patients With Controlled Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCOX189A2475
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Osteoarthritis With Controlled Hypertension
Keywords: Osteoarthritis, controlled hypertension, lumiracoxib, ibuprofen, high blood pressure
MeSH Terms: conditions — Osteoarthritis; Hypertension | interventions — lumiracoxib

INTERVENTIONS:
Drug: Lumiracoxib

SUMMARY:
This randomized study will compare the effect of lumiracoxib, ibuprofen and placebo on 24-hour blood pressure profile and on urinary excretions of eicosanoids in controlled hypertensive patients who have osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients of at least 50 years of age.
* Female patients must be either post-menopausal for one year, surgically sterile, or using effective contraceptive methods such as barrier method with spermicide or intra-uterine device. Oral contraceptives use is not allowed 4 weeks prior screening and throughout the duration of the study. Patients on hormonal replacement therapy are allowed if they have been on a stable dose for at least 6 months.
* Primary osteoarthritis of the hand, hip or knee according to American College of Rheumatology (ACR) criteria or osteoarthritis of the spine. One joint will be identified as the target joint and will be evaluated throughout the duration of the trial.
* Is expected to need non-steroidal anti-inflammatory drugs (NSAID) or simple analgesic therapy for osteoarthritis for at least the next 6 weeks.
* Controlled hypertension with mean sitting systolic blood pressure (MSSBP) <140 mmHg and mean sitting diastolic blood pressure (MSDBP) <90 mmHg (mean of 3 cuff blood pressure measurements). Patients must have taken the same fixed dose of antihypertensive medication(s) on a regular basis for at least 3 consecutive months prior to screening and are not expected to adjust their antihypertensive medication(s) during the study. Regular wake-up times which are expected to continue for the duration of the trial.

Exclusion Criteria:

* History of hypersensitivity to any of the study drugs or to drugs with similar chemical structures.
* Patients who have any known allergic-type reactions after taking acetylsalicylic acid or NSAIDs which may include (but are not limited to) history of asthma, acute rhinitis, nasal polyps, angioneurotic edema, urticaria or other allergic-type reactions
* History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/ml).
* History of cardiac and cerebral thrombotic/ ischemic diseases and/ or events as listed below:

angina pectoris (of any severity) or other evidence of coronary heart disease; myocardial infarction; coronary heart disease with ECG-evidence of silent myocardial infarction; coronary artery bypass grafting (CABG) or percutaneous coronary intervention (any PCI procedure); clinically significant carotid artery stenosis or history of carotid endarterectomy; congestive heart failure, NYHA class II - IV; second or third degree heart block in the absence of permanent pacing and all potentially life-threatening arrhythmia or symptomatic arrhythmia; clinically significant valvular heart disease; cerebrovascular disease; peripheral arterial disease

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2006-11; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in average 24-hour systolic blood pressure (BP) derived from ambulatory blood pressure monitoring (ABPM) after 4 weeks of treatment
Urinary eicosanoid excretion

SECONDARY OUTCOMES:
Change from baseline in average 24-hour diastolic BP derived from ABPM after 4 weeks of treatment
Day and night time blood pressure (systolic and diastolic) derived from ABPM after 4 weeks of treatment
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis, East Hanover, New Jersey, United States